CLINICAL TRIAL: NCT02523664
Title: Why Does Cortisol Enhance Memory Retrieval in Patients With Borderline Personality Disorder and Posttraumatic Stress Disorder? Investigating the Neuronal Correlates of Cortisol Administration and the Effects of Stress Exposure
Brief Title: Neural Correlates of Stress Hormones
Acronym: Cort-fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: WI-3396-2
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Borderline Personality Disorder; PTSD
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone (Active Comparator): 10 mg hydrocortisone orally
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — effects of hydrocortisone on memory while fMRI
  Arms: Hydrocortisone
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate which neuronal correlates underlie cortisol-induced enhancement of memory retrieval in PTSD and BPD.

DETAILED DESCRIPTION:
The investigators have recently shown that hydrocortisone enhances rather than impairs memory retrieval in patients with posttraumatic stress disorder (PTSD) and borderline personality disorder (BPD). In contrast, in healthy participants memory retrieval was impaired after hydrocortisone compared to placebo.

The proposed studies aim to further investigate these findings and to understand the underlying neuronal correlates. Thus, the mechanisms of enhanced memory retrieval after hydrocortisone in patients with BPD and PTSD will be investigated by fMRI.

In a placebo-controlled study, the effects of 10mg hydrocortisone on brain activity, in particular the hippocampus, will be investigated in patients with PTSD and BPD and will be compared with those in healthy control participants. During the fMRI session, a declarative memory task (retrieval of a previous learned word list) and an autobiographical memory test will be performed. Effects of hydrocortisone on resting state brain activity and the neuronal correlates of memory retrieval will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Borderline Personality Disorder
* Clinical diagnosis of PTSD
* females without psychiatric disorders as control group
* right handed

Exclusion Criteria:

* fMRI exclusion criteria e.g. metal implants, pregnancy, left-handedness, and claustrophobia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
brain activation after hydrocortisone | 20 min
  fMRI

SECONDARY OUTCOMES:
memory retrieval after hydrocortisone | 10 minutes
  Retrieval of a previous learned word list
memory retrieval after hydrocortisone | 20 minutes
  autobiographic memory retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany